CLINICAL TRIAL: NCT05866458
Title: Radiation OmisSion in PAtients With CLinically Node Negative Breast Cancer Undergoing Lumpectomy and With a PathologIc Complete REsponse After Neoadjuvant Chemotherapy
Brief Title: Radiation OmisSion in PAtients With CLinically Node Negative Breast Cancer Undergoing Lumpectomy
Acronym: ROSALIE
Status: Recruiting | Type: Observational
Sponsor: Ontario Clinical Oncology Group (OCOG) (Other)
Responsible Party: Sponsor
Other Study IDs: OCOG-2022-ROSALIE
Record Dates: First submitted 2023-05-10; First posted 2023-05-19 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
Keywords: Clinically node negative breast cancer; Ipsilateral breast tumour recurrence; Neoadjuvant chemotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single Arm Cohort: The study population consists of women with newly diagnosed T1-3 node negative breast cancer with no clinical evidence of distant metastatic disease, that have been treated with NAC, BCS and axillary staging surgery with final pathology demonstrating a pCR (defined as absence of residual invasive and in situ breast cancer within the breast or lymph nodes).

SUMMARY:
To de-escalate radiation therapy in women with breast cancer.

DETAILED DESCRIPTION:
The study is a prospective, multi-center, single arm cohort study of omission of adjuvant whole breast radiation therapy (WBRT) following breast conserving surgery (BCS) in patients with a pathological complete response (pCR) following neoadjuvant chemotherapy (NAC). Eligible and consenting female patients with newly diagnosed T1-3 node negative breast cancer with no clinical evidence of distant metastatic disease, who have been treated with NAC, BCS and axillary staging surgery with final pathology demonstrating a pCR (ypT0N0) will be enrolled to the study and followed. The first analysis is planned when follow-up is a median of 5 years. Study participants will not receive adjuvant WBRT, the current standard of care.

The primary outcome is ipsilateral breast tumour recurrence (IBTR) at median 5-year follow-up. Study participants will be followed and assessed for local recurrence, regional recurrence, distant recurrence, DFS and OS. In addition, any additional breast cancer treatments received by the participant for the first recurrence event including repeat BCS, mastectomy, additional systemic therapy and radiation therapy (RT) will be documented. The planned sample size is 352 study participants.

ELIGIBILITY:
Inclusion Criteria:

1. Female patient with a new histological diagnosis of clinical T1-3 N0 breast cancer (any tumour sub-type).
2. Negative lymph node involvement at initial presentation, documented by imaging (US or MRI), fine needle aspiration (FNA) or core needle biopsy.
3. Treated with a minimum of 8 weeks NAC, with patients with Her2+ disease receiving targeted anti-Her2+ therapy.
4. Marker clip placed in the tumour bed prior to or during neoadjuvant chemotherapy when the tumour can still be identified.
5. Treated by BCS with complete excision of the tumour bed and axillary staging surgery (either sentinel lymph node biopsy or axillary lymph node dissection).
6. Final pathology demonstrating a pCR [defined as absence of residual invasive and in-situ breast cancer within the breast or lymph nodes (ypT0N0)].

Exclusion Criteria:

1. Age less than 50 years.
2. Inflammatory breast cancer or breast cancer invading the skin or chest wall (T4 disease).
3. Multicentric disease (i.e., breast cancer involving more than one quadrant in the same breast).
4. Prior history of ipsilateral or contralateral in-situ or invasive breast cancer. Patients with a history of lobular carcinoma in-situ (LCIS) are ineligible.
5. Synchronous contralateral in-situ or invasive breast cancer.
6. BRCA (breast cancer gene) 1 or 2 genetic mutation carrier, or other genetic mutation present associated with increased risk of breast cancer.
7. Other previous non-breast malignancies except adequately treated non-melanoma skin cancers, in situ cancers or other cancers curatively treated with no evidence of disease for ≥ 5 years.
8. Inability to complete entire course of neoadjuvant therapy (minimum of 8 weeks of treatment).
9. Patients with HR+ (hormone receptor) disease who are not planned to have endocrine therapy initiated.
10. Patients with Her2+ disease who have not received or are not planned to receive Her2 targeted therapy.
11. ECOG (Eastern Cooperative Oncology Group) performance status > 3.
12. Inability to provide informed consent.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Written informed consent will be obtained from all eligible patients who agree to participate. Until the patient has been completely informed of the study, has freely consented to take part in the study and has signed and dated an informed consent form that has received documented approval by an authorized Research Ethics Board (REB), no study related assessments, including those required for screening can be performed.
Sampling Method: Non-Probability Sample
Enrollment: 352 (Estimated)
Dates: Start 2024-03-12 (Actual); Primary Completion 2031-10 (Estimated); Study Completion 2031-10 (Estimated)

PRIMARY OUTCOMES:
Ipsilateral breast tumour recurrence (IBTR) | 5 years
  defined as ipsilateral recurrence (invasive or insitu) in the ipsilateral breast or chest wall. Histological evidence of IBTR is required. All such events will be reviewed by a central adjudication committee.

SECONDARY OUTCOMES:
Mastectomy free interval | 5 years
  defined as time from registration to undergoing ipsilateral mastectomy.
Relapse free interval (RFI) | 5 years
  defined as time from registration to recurrence of invasive disease in the ipsilateral breast, regional nodes (axilla, supraclavicular, or internal mammary), distant areas beyond local or regional limits (distant recurrence), and death from breast cancer.
Disease free survival (DFS) | 5 years
  defined as time from registration to in breast invasive tumour recurrence, regional invasive recurrence, distant recurrence, contralateral breast cancer, second primary non-breast cancers, death from breast cancer, and death from non-breast cancer.
Overall survival (OS) | 5 years
  defined as time from registration to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Elena Parvez, MD, Principal Investigator — Juravinski Cancer Centre; Thierry Muanza, MD, Principal Investigator — Jewish General Hospital; Mark Basik, MD, Principal Investigator — Jewish General Hospital
Locations (12):
- Canada (12):
  - BC Cancer - Centre for the North, Prince George, British Columbia
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston, Kingston, Ontario
  - Thunder Bay Regional Health Sciences Centre, Thunder Bay, Ontario
  - Sunnybrook Health Sciences -Odette Cancer Centre, Toronto, Ontario
  - CHUM - Centre Hospitalier de L'Université de Montréal, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - CHU de Quebec - Universite Laval, Québec, Quebec
  - Centre hospitalier de Lanaudière, Saint-Charles-Borromée, Quebec
  - Centre Hospitalier Trois Rivieres Ste-Marie, Trois-Rivières, Quebec
  - McGill University Health Centre (MUHC), Montreal, Q

IPD SHARING:
Plan to Share IPD: No